CLINICAL TRIAL: NCT06236620
Title: Zinc Absorption in Flakes Derived from Sprouted or Hydrothermally Processed Wheat
Acronym: Wheatflakes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Professor, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: S64419
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Zinc Absorption
Keywords: zinc absorption; zinc bio-availability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control wheat flakes (Active Comparator): Wheat flakes made of whole derived from unprocessed wheat
  Interventions: Dietary Supplement: Processing of wheat
- Flakes from sprouted wheat (Active Comparator): Wheat flakes made of whole derived from sprouted wheat
  Interventions: Dietary Supplement: Processing of wheat
- Flakes from hydrothermally processed wheat (Active Comparator): Wheat flakes made of whole derived from hydrothermally processed wheat
  Interventions: Dietary Supplement: Processing of wheat

INTERVENTIONS:
Dietary Supplement: Processing of wheat — Investigating if the consumption of sprouted or hydrothermally processed wheat affects the iron and zinc absorption in humans

SUMMARY:
The aim of this project is to investigate whether the increased zinc bio-accessibility values in sprouted or hydrothermally processed wheat is reflected in an increased zinc absorption in human subjects after consuming breakfast flakes derived from such processed wheats.

DETAILED DESCRIPTION:
The zinc study is a randomised crossover design with two different meals (control wheat flakes and flakes derived from sprouted wheat or flakes derived from hydrothermally processed wheat) spiked with a specific zinc isotope. The study contains two test groups (I and II) of 26 and 10 participants, respectively. Both test groups will consume the control wheat flakes, whereas test group I will consume the flakes from sprouted wheat and group II the flakes from hydrothermally processed wheat randomised over two test days. An intravenous dose of Zn will be given on day 1 of the study and the zinc isotope composition in the urine of the participants will be measured on day 1,5,6,7 and 8 of the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI range 18.5-25.0 kg/m²
* Regular diet with 3 meals a day (at least 5 times a week)

Exclusion Criteria:

* Intake of vitamin and/or mineral supplements during and 2 weeks before the stud
* Intake of antibiotics 3 months prior to the study
* Intake of medicines that have an impact on the gastrointestinal tract during and 2 weeks before the study
* Previous or current gastrointestinal (e.g. Crohn's disease), endocrine or eating disorders or other gastrointestinal history
* Previous or current substance/alcohol dependence or abuse (> 2 units per day/14 units per week)
* Currently smoking (have smoked in the last 28 days) or willingness to smoke during the study period
* Pregnant or lactating or wishing to become pregnant in the period of the study
* Allergy or intolerance to wheat (coeliac disease, gluten sensitivity) or citric acid
* Adherence to vegan or vegetarian diets or special diets (weight loss, gluten-free etc…)
* Blood donation in the 6 months prior to the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Zinc absorption | day 1 (before test meal) and day 5,6,7 and 8
  Zinc isotope abundance in urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, Prof., Principal Investigator — KU Leuven
Locations (1):
- KU Leuven/UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No